CLINICAL TRIAL: NCT02956135
Title: Relationship Between Dysfunctions of Movement in the Lower Back and Pelvis With Overuse Injuries in Handball Players
Status: Completed | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Fco. Javier Montanez Aguilera, PhD, Cardenal Herrera University
Other Study IDs: CEU C Herrera
Record Dates: First submitted 2016-11-01; First posted 2016-11-07 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-11

CONDITIONS: Dysfunction;Joint; Overuse Injury
MeSH Terms: conditions — Joint Diseases; Cumulative Trauma Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to assess the relationship between the presence of overuse injuries and failure to control of movement in those areas. For this, participants will perform some tests related to movement dysfunction lumbar-pelvic area to check for faults in one or more movement planes.

DETAILED DESCRIPTION:
Handball is considered a high intensity sport even though the 70% of the time the game is standing or walking. The large number of repetitions of high intensity activities such as sprinting or jumping, associated with physical contact with opposing players, make this sport in a physically demanding activity. Furthermore, overuse injuries have been widely described but poorly quantified. In addition, is necessary to know the influence of static lumbar-pelvic position in low back pain and its correlation with stability. Not only strength is important for a good quality of movement, there should also be a specific muscle activation in order for a correct motor pattern. This coordinated action must be I just by the action of muscles agonists, antagonists and synergists.The aim of this study is to assess the relationship between the presence of overuse injuries and failure to control of movement in those areas. For this, participants will perform some tests related to movement dysfunction lumbar-pelvic area to check for faults in one or more movement planes.

ELIGIBILITY:
Inclusion Criteria:

* Players from the first team
* Without injury that does not allow movement tests

Exclusion Criteria:

* Spinal cord injury or tumor, myelopathy, neuropathy and spondylitis and spondylolisthesis in the lumbar spine.
* Tumors or major injuries in the knee or hip.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Fertiberia Puerto de Sagunto Club handball players, from national first division of Spain
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Control of lumbopelvic movement | Once, at baseline
  It is seven tests to check the control of lumbopelvic movement. They are low-intensity tests to assess the ability to control movement of the stabilizing musculature. The mobilizing muscles should not have a dominant role in these tests. The test were recorder on video to be analyzed later

SECONDARY OUTCOMES:
Pain sensation | Once, at baseline
  Pain sensation measured with a visual analog scale
Epidemiological registry | Through study completion, an average of 2 year
  Information related to injuries suffered by players

CONTACTS AND LOCATIONS:
Overall Officials: F Javier Montañez-Aguilera, PhD, Study Director — CEU Cardenal Herrera University
Locations (1):
- F Javier Montañez-Aguilera, Moncada, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karcher C, Buchheit M. On-court demands of elite handball, with special reference to playing positions. Sports Med. 2014 Jun;44(6):797-814. doi: 10.1007/s40279-014-0164-z. PMID 24682948
- [Background] Michalsik LB, Aagaard P, Madsen K. Locomotion characteristics and match-induced impairments in physical performance in male elite team handball players. Int J Sports Med. 2013 Jul;34(7):590-9. doi: 10.1055/s-0032-1329989. Epub 2012 Dec 20. PMID 23258606
- [Background] Bere T, Alonso JM, Wangensteen A, Bakken A, Eirale C, Dijkstra HP, Ahmed H, Bahr R, Popovic N. Injury and illness surveillance during the 24th Men's Handball World Championship 2015 in Qatar. Br J Sports Med. 2015 Sep;49(17):1151-6. doi: 10.1136/bjsports-2015-094972. Epub 2015 Jul 17. PMID 26282368
- [Background] Danis CG, Krebs DE, Gill-Body KM, Sahrmann S. Relationship between standing posture and stability. Phys Ther. 1998 May;78(5):502-17. doi: 10.1093/ptj/78.5.502. PMID 9597064
- [Background] Van Dillen LR, Sahrmann SA, Norton BJ, Caldwell CA, Fleming DA, McDonnell MK, Woolsey NB. Reliability of physical examination items used for classification of patients with low back pain. Phys Ther. 1998 Sep;78(9):979-88. doi: 10.1093/ptj/78.9.979. PMID 9736895
- [Background] Comerford MJ, Mottram SL. Movement and stability dysfunction--contemporary developments. Man Ther. 2001 Feb;6(1):15-26. doi: 10.1054/math.2000.0388. PMID 11243905